CLINICAL TRIAL: NCT06701799
Title: CAF in Association with Different Thickness of L-PRF Membranes of for the Treatment of RT1 Gingival Recession: a Randomized Controlled Clinical Trial.
Brief Title: Clinical Evaluation of Gingival Biotype Changes Using a Coronally Advanced Flap (CAF) in Combination with Leucocyte and Platelet- Rich Fibrin (L-PRF) Membranes of Different Thickness for the Treatment of RT1 Gingival Recession: a Randomized Controlled Clinical Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 211124
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Mucogingival Defects; Recession, Gingival; Gingival Recession, Mucogingival Surgery; L-PRF
Keywords: Coronally Advanced Flap; L-PRF; Platelet concentrate; Gingival Recession; Gingival Biotype
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAF+ L-PRF 2 mm (Experimental): Coronally Advanced Flap combined with in combination with a membrane 2 mm in thickness of L-PRF for the Treatment of RT1 Gingival Recession.
  Interventions: Procedure: CAF+ L-PRF 2 mm
- CAF+ L-PRF 1 mm (Experimental): Coronally Advanced Flap combined with in combination with a membrane 1 mm in thickness of L-PRF for the Treatment of RT1 Gingival Recession.
  Interventions: Procedure: CAF+ L-PRF 1 mm

INTERVENTIONS:
Procedure: CAF+ L-PRF 1 mm — The extent of the depth of the recession will be reported on the anatomical papillae and, after adding 1 mm, 2 horizontal incisions of approximately 3 mm will be made at the base of the surgical papillae laterally to the recession.Two divergent releasing incisions will be made extending approximately 2-3 mm into the alveolar mucosa.The surgical papillae will be detached in partial thickness. A full thickness dissection will be performed from the bottom of the recession to expose approximately 3mm of the crest bone.A partial thickness dissection will be performed in the most apical portion of the flap until complete passivation of the flap is obtained. The L-PRF membrane 1 mm in thickness, will be positioned at the level of the de-epithelialised anatomical papillae.The flap will be repositioned coronally suturing the anatomical papillae on the surgical ones, using a Non-Resorbable 5.0 Polyamide Suture.
  Arms: CAF+ L-PRF 1 mm
Procedure: CAF+ L-PRF 2 mm — The extent of the depth of the recession will be reported on the anatomical papillae and, after adding 1 mm, 2 horizontal incisions of approximately 3 mm will be made at the base of the surgical papillae laterally to the recession.Two divergent releasing incisions will be made extending approximately 2-3 mm into the alveolar mucosa.The surgical papillae will be detached in partial thickness. A full thickness dissection will be performed from the bottom of the recession to expose approximately 3mm of the crest bone.A partial thickness dissection will be performed in the most apical portion of the flap until complete passivation of the flap is obtained. The L-PRF membrane 2 mm in thickness, will be positioned at the level of the de-epithelialised anatomical papillae.The flap will be repositioned coronally suturing the anatomical papillae on the surgical ones, using a Non-Resorbable 5.0 Polyamide Suture.
  Arms: CAF+ L-PRF 2 mm

SUMMARY:
Gingival thickness plays a key role not only in the etiology but also in the treatment of gingival recessions. More recently, authors reported that as the gingival thickness decreases, the gingival recession severity increases . When gingival inflammation occurs, if the tissue is thin the consequent destruction can quickly produce a gingival recession (GR) .

When treating a gingival recession, the clinician should aim not only to completely cover the exposed root surface but also to prevent a future recession recurrence. The treatment gold standard is the CAF associated with connective tissue graft. This technique has demonstrated high rates in gingival recession reduction and positive predictability in obtaining complete root coverage. However, some disadvantages about this surgical approach can be easily highlighted: patients experience more discomfort, longer chair-time it's necessary and a second wound area is created. In this scenario, The Platelet rich in fibrin and leucocyte (L-PRF) could be a valuable alternative treatment of gingival defects. It's a platelet concentrate, obtained by a fast and simple procedure that does not require anticoagulant and bovine thrombin. It can also be categorized as a live tissue thanks to platelets, leukocytes, growth factors and stem cells trapped in a polymerized fibrin mesh. L- PRF is used in various fields of regenerative medicine; It promotes stabilization and revascularization of the flaps, contributes to soft tissue wound healing and reduces post-operative discomfort. The purpose of this study will be to evaluate if the different thickness of platelet- rich fibrin (L-PRF) membranes in association with a Coronally Advanced Flap (CAF), for the treatment of RT1 gingival recessions, may influence the Complete Root Coverage (CRC).

DETAILED DESCRIPTION:
This prospective, randomized and controlled clinical trial will compare: CAF +1 mm thick L-PRF membrane versus CAF +2 mm thick L-PRF membrane for the treatment of RT1 gingival recession. From each patient a single recession on a single tooth will be selected. Clinical parameters will be evaluated at base-line and after 6 months.

The protocol is approved by the "G. D'Annunzio" University Ethical Committee. This study is in accordance with the Declaration of Helsinki of 1975. Patients will be recruited from the Unit of Periodontology, "G. D'Annunzio" University of Chieti-Pescara, Italy. All the volunteer candidates will sign a written informed consent.

The trial director will be responsible for randomly assigning patients to treatment after enrollment and will not involve with the clinical interventions or the study measurements. A computer-generated table will be used to make the random assignment, known only to the trial director. An opaque envelope will conceal group allocation and will be opened just before the intervention surgery. Matching between group and treatment will be performed by a figure extraneous to the experimentation, responsible even for keeping and breaking the blinding, and known only to him.

Patients and examiners will be masked to group membership; clinical examiners will be blinded to each other. The study analyst will be also blind to group membership. The analyst will receive the data by groups labeled as A and B. The blind will not be broken until after study completion. Complete root coverage (CRC) will be assumed as the main outcome at 6 months after treatment. At baseline and 6 months after surgery, the following clinical measurements will be also recorded on the mid-buccal point of exposed root surface: Gingival thickness (GT) will be determined using a stent at a mid-buccal location about 1 mm apical to the pocket depth (PD) level with a #15 endodontic reamer with a silicon disk stop. The soft tissue will be gently pierced at a 90° angle, until hard tissue will be felt. Once the silicon disk will be in contact with the soft tissue surface, it will be fixed by a drop of cyanoacrylate adhesive. After the careful removal of the reamer, the distance between the reamer tip and the stop will be measured with a calliper accurate to the nearest 0.1 mm. The other measurements will be taken with a periodontal probe and will be recorded to the nearest millimetre as follows: Gingival recession (GR) will be measured as the distance from the cement-enamel junction (CEJ) to the mid-buccal point of the gingival margin. PD and Clinical attachment level (CAL) will be measured as the distance between the bottom of the pocket and the gingival margin and CEJ, respectively. Keratinized tissue (KT) will be recorded from the mid-buccal point of the gingival margin to the mucogingival junction. Root coverage esthetic score (RES) (Cairo et al., 2009) will be used for assessing aesthetic outcomes of root coverage procedures. PROMs will also be evaluated. The degree of general discomfort (D) experienced will be assessed on a VAS scale (0-10). Patient-reported aesthetic satisfaction (PRES) at T1 will also be quantified on a VAS scale (0-10). Overall treatment satisfaction (OTS) at T1 will be assessed by asking each patient if they would undergo surgery again (yes/no). Thirty ml of blood samples will be collected in 10-ml tubes without anticoagulant and promptly centrifuged at 3,000 revolutions per minute for 10 minutes. The L-PRF membranes will be realized by a standardized compression of the clot for 120 seconds with 130 grams; the membranes will be put one on each other till obtaining a resultant membrane of the desired thickness: 1 or 2 mm. Exposed and intrasulcular root surface will be accurately scaled using curettes. A coronally advanced flap technique (CAF) will be used to treat the recession defect. The ﬂap will be elevated as follows: an intrasulcular incision will be performed around the selected tooth, the incision moves on contiguous papillae area, avoiding the gingival margin of adjacent teeth. From each side, from coronal to apical, an oblique incision will be carried out. A split-full-split dissection will be undertaken until the CEJ could be passively cover by the flap. Both papillae will be de-epithelialized. The 1 mm L-PRF membrane will be be placed over the exposed root surface of the CAF+ L-PRF 1mm group and the 2 mm L-PRF membrane in the CAF+ L-PRF 2 mm group. The gingival defect will be fully lined by grafts that mildly cover the neighbouring sub-papillae areas. In each group, ﬂap will be coronally positioned and sutured over the enamel in a tension-free position.

All patients will receive 2 g/day amoxicillin+clavulanic acid for 6 days for post-operative infection prevention; 400 mg of oral ibuprofen, twice daily, will control the pain; 0.12% chlorhexidine rinses, twice daily for 3 weeks, will be prescribe to the patients. Sutures will be removed after 14 days. Only 2-4 weeks after sutures removal, respectively, cautious brushing by a soft toothbrush and interdental brushing will be recommend; meantime, the patients use a 1% chlorhexidine gel twice daily. Weekly supra-gingival professional hygiene and motivational reinforcement will be administer to the patients for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Systemic factors (no systemic diseases; no coagulation disorders; no medications affecting periodontal status in the previous 6 months; no pregnancy or lactation)
* Never smokers/former smokers >=10years
* Full-mouth plaque score (FMPS)and a full-mouth bleeding score (FMBS) lower than 15%
* No periodontal surgery on the experimental sites
* >= 20 teeth without mobility
* No presence of cervical carious lesions or periapical lesions at experimental sites
* At least one RT1 buccal gingival recession

Exclusion Criteria:

* Systemic diseases
* Coagulation disorders
* Medications affecting periodontal status in the previous 6 months
* Pregnancy or lactation
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  Percentage of experimental sites that achieved complete root surface coverage.

SECONDARY OUTCOMES:
Keratinized tissue width | 6 months
  Distance between gingival margin and Mucogingival Junction.
Clinical attachment level | 6 months
  Distance between cementoenamel junction(CEJ) and depth of the pocket.
Gingival Recession | 6 months
  Distance from cementoenamel junction and gingival margin.
Gingival thickness | 6 months
  Gingival tissue thickness evaluated 2 mm apical to the recession.
Pocket depth | 6 months
  Distance between gingival margin and bottom of the pocket.
Discomfort | 4 weeks
  Evaluation of post-operative discomfort using Visual Analogue Scale (VAS).The scale is represented by a straight horizontal line of fixed length, generally 10 cm. Extremities are defined as extreme limits of the parameter to be measured, oriented from left (worst) to right (best).
Patient-Reported Esthetic Satisfaction | 6 months
  Patient-reported esthetic satisfaction (PRES) quantified on a VAS scale (0-10), will be recorded after observing simultaneously 2 standardized photographs showing the treated site +2 mesial and 2 distal teeth and the MGJ.
Root Coverage Esthetic Score | 6 months
  This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Innovative Technologies in Medicine and Dentistry, Chieti, Chieti, CH, Italy